CLINICAL TRIAL: NCT04905667
Title: A Single Center, Randomized, Blind, Parallel Controlled, Single Dose Pharmacokinetic Study of Recombinant Humanized Anti-HER-2 Monoclonal Antibody Injection GB221 in Comparison With Herceptin ® in Chinese Healthy Adult Volunteers
Brief Title: Single Dose Pharmacokinetic Study of GB221 in Comparison With Herceptin ®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 221-005
Record Dates: First submitted 2021-03-02; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Pharmacokinetics; anti-HER-2 human monoclonal antibody; Herceptin; GB221
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blind (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GB221 group (Experimental): 6 mg/kg, single dose, intravenous infusion, 90-100 min
  Interventions: Drug: GB221
- Herceptin group (Active Comparator): 6 mg/kg, single dose, intravenous infusion, 90-100 min
  Interventions: Drug: Herceptin

INTERVENTIONS:
Drug: GB221 — 6 mg/kg, single dose, intravenous infusion, 90-100 min
  Arms: GB221 group
Drug: Herceptin — 6 mg/kg, single dose, intravenous infusion, 90-100 min
  Arms: Herceptin group

SUMMARY:
This is a single center, randomized, blind, parallel controlled clinical trial. The primary objective is to evaluate the single dose pharmacokinetics of recombinant Humanized anti-HER-2 monoclonal antibody injection GB221 in comparison with Herceptin ® in Chinese healthy adult volunteers. The main aim is to study the pharmacokinetic similarity between GB221 and Herceptin ®.

DETAILED DESCRIPTION:
Subjects will enroll in random order, and be divided into two groups, then receive a single dose (6 mg/kg) of GB221 or Herceptin ®, and accept observation for 42 days. Throughout the course, safety data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed informed consent form;
* 2. Healthy adult volunteers aged between 18 and 45, male or female;
* 3. Medical examination as required within 28 days, body mass index (BMI) 19.0 ~ 24.0, weight≥50 kg for men, ≥45 kg for women, and≤ 75 kg for both;
* 4. Agreed with taking reliable contraceptive measures, and no fertility planning from the beginning to the end of the study within 6 months;
* 5.Subject can communicate well with the investigators and complete the study according to the study regulations.

Exclusion Criteria:

* 1. Pregnant or lactating women, or positive in either blood or urine pregnancy test; or unwilling to take effective contraceptive measures during the trial and within 6 months after the end of the trial at fertile age;
* 2. Allergic constitution; or history of allergic to experimental drug ingredient or any drug or food or pollen; or abnormal serum immunoglobulin E (IgE) test;
* 3. History of drug abuse, or positive urine test for drug;
* 4. History of the central nervous system, cardiovascular system, kidney, liver, digestive system, respiratory system, metabolic system or other significant diseases. History of high blood pressure, or clinically significant systolic blood pressure≥140 mmHg/diastolic blood pressure≥90 mmHg;
* 5. Family history of cancer, or tumor markers (male: CEA, AFP, PSA, CA-125; Female: CEA, AFP, CA-153, CA-125) positive.
* 6. Participated in other clinical trials of drug or used drugs harmful to major organs within 3 months;
* 7. Blood donation within 3 months;
* 8. Used prescription or OTC drugs within 14 days;
* 9. Left ventricular ejection fraction (LVEF) < 60%;
* 10. ALT or AST > 1.5 ULN, Cr > ULN;
* 11. WBC < 0.8 LLN or > 1.2 ULN; ANC < 0.8 LLN; PLT < 0.8 LLN; HGB < 0.9LLN.
* 12. HBs-Ag, HCV-Ab, anti-HIV or TP-Ab positive;
* 13. Anti-drug antibody (ADA) test positive;
* 14.History of psychosis;
* 15. History of postural hypotension;
* 16. More than 5 cigarettes per day;
* 17. More than 28 units of alcohol per week; Or alcohol breath test positive within 24 hours before pre-dose;
* 18. History of dizziness of blood or needle;
* 19. Unsuitable for other reasons.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
AUC0-t | Day 43
  compare the pharmacokinetic AUC0-t parameters of GB221 and Herceptin ®
AUC0-∞ | Day 43
  compare the pharmacokinetic AUC0-∞parameters of GB221 and Herceptin ®
Cmax | Day 43
  compare the pharmacokinetic Cmax parameters of GB221 and Herceptin ®

SECONDARY OUTCOMES:
Tmax | Day 43
  compare the pharmacokinetic Tmax parameters of GB221 and Herceptin ®
t1/2 | Day 43
  compare the pharmacokinetic t1/2 parameters of GB221 and Herceptin ®
CL | Day 43
  compare the pharmacokinetic CL parameters of GB221 and Herceptin ®
Vd | Day 43
  compare the pharmacokinetic Vd parameters of GB221 and Herceptin ®
Ke | Day 43
  compare the pharmacokinetic Ke parameters of GB221 and Herceptin ®
ADA | Day 43
  compare the incidence of ADA in of GB221 and Herceptin ® group
Nab | Day 43
  compare the incidence of Nab in of GB221 and Herceptin ® group

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No